CLINICAL TRIAL: NCT02656277
Title: Efficacy of First Time Anterior Shoulder Decision Tool in a Randomized Control Trial
Brief Title: Efficacy of First Time Anterior Shoulder Decision Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00066738
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision tool (Experimental): The decision tool includes a questionnaire and statistical model used to determine how patient preference regarding shoulder pain, physical limitations, physical therapy, recovery period, prognosis, and cost impact choice of surgical versus non-surgical intervention.
  Interventions: Other: Decision Tool
- Information on Shoulder Dislocation (Active Comparator): Subjects in this arm will receive the standard of care information available to patients to make this treatment decision.
  Interventions: Other: Information on Shoulder Dislocation

INTERVENTIONS:
Other: Decision Tool
  Arms: Decision tool
Other: Information on Shoulder Dislocation
  Arms: Information on Shoulder Dislocation

SUMMARY:
This study is a randomized controlled trial using Duke patients to test, compared to the standard of care, a questionnaire and statistical model used to determine how patient preference regarding shoulder pain, physical limitations, physical therapy, recovery period, prognosis, and cost impact choice of surgical versus non-surgical intervention.

Phase 1 of this study is the initial testing of the instrument and involves a small group of up to 10 individuals who will partake in one-on-one interviews while completing the Shoulder Injury Survey to provide feedback. In Phase 2 of this study, 200 subjects will be randomized to receive either the Decision Tool or the standard Information on Shoulder Dislocation

DETAILED DESCRIPTION:
An anterior shoulder dislocation is a common problem for people between the ages of 15 to 35. Recurrent instability is common and dependent on age and gender. Treatment options include surgical intervention and repair or non-surgical options that include intensive rehabilitation. Level I evidence suggests early surgical repair can significantly reduce the risk of recurrent instability. The risk of arthritis is increased with multiple dislocation episodes.

Traditionally, the combination of 1) history and physical exam performed by the provider, 2) clinical and diagnostic tools to assess the extent of injury and impact on physical activity, and 3) patient-voiced preference has guided the selection of an optimal solution for an individual patient. When providing a recommendation to individual patients and their unique circumstances, the health care provider may gather patient preferences on factors such as desire to avoid pain, chance of recurrent shoulder dislocation, time needed for rehabilitation and physical therapy, and operative versus non-operative costs. Surgical and non-surgical options have distinct differences in these outcomes. When combined, the interaction between these variables creates important tradeoffs of risks and benefits for each option.

No studies have been conducted to determine the objective weight of these different dimensions of patient preferences and how they might guide the provider-patient conversation. Conjoint analysis is a statistical method that seeks to quantify the relative importance of various aspects of the decision-making process, such as cost or probability of repeat injury as described above. Combined with a validated survey tool, conjoint analysis of patient preferences in shoulder repair can assist the physician in recommending a patient-centered option.

ELIGIBILITY:
Inclusion Criteria:

- Shoulder dislocation

Exclusion Criteria:

* Prior surgery for shoulder stabilization
* Inability to complete enrollment forms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Preference Survey | 2 months
  patient-voiced preferences guiding solution

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mather, MD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hutyra CA, Smiley S, Taylor DC, Orlando LA, Mather RC 3rd. Efficacy of a Preference-Based Decision Tool on Treatment Decisions for a First-Time Anterior Shoulder Dislocation: A Randomized Controlled Trial of At-Risk Patients. Med Decis Making. 2019 Apr;39(3):253-263. doi: 10.1177/0272989X19832915. Epub 2019 Mar 5. PMID 30834817